CLINICAL TRIAL: NCT05656495
Title: An Open Randomized Multicenter Comparative Study to Evaluate the Efficacy, Safety and Tolerability of the Use of Ambervin® for Intramuscular Administration and for Inhalation in Patients Hospitalized With COVID-19
Brief Title: Efficacy and Safety of Ambervin® and Standard Therapy in Hospitalized Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Promomed, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMB-112021
Record Dates: First submitted 2022-12-15; First posted 2022-12-19 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Ambervin
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ambervin intramuscularly (Experimental): Arm 1 (n=104) receives the study drug Ambervin for intramuscularly administration 1 mg 1 time per day. The course of treatment is 10 days.
  Interventions: Drug: Tyrosyl-D-alanyl-glycyl-phenylalanyl-leucyl-arginine succinate intramuscularly
- Ambervin inhaled (Experimental): Arm 2 (n=105) receives the study drug Ambervin for inhalation administration 10 mg 1 time per day. The course of treatment is 10 days.
  Interventions: Drug: Tyrosyl-D-alanyl-glycyl-phenylalanyl-leucyl-arginine succinate inhaled
- Standard of care (Active Comparator): Arm 3 (n=104) patients receive standard therapy prescribed in accordance with the recommended treatment regimens included in the InterimGuidelines for the prevention, diagnosis and treatment of new coronavirus infection (COVID-19) approved by the Russian Ministry of Health by decision of the investigator and taking into account the availability of drugs at the study site
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Tyrosyl-D-alanyl-glycyl-phenylalanyl-leucyl-arginine succinate intramuscularly — lyophilizate for preparation of solution for intramuscular administration 1 mg 1 time per day for 10 days
  Other Names: Ambervin intramuscularly
  Arms: Ambervin intramuscularly
Drug: Tyrosyl-D-alanyl-glycyl-phenylalanyl-leucyl-arginine succinate inhaled — lyophilizate for preparation of solution for inhalation administration 10 mg 1 time per day for 10 days
  Other Names: Ambervin inhaled
  Arms: Ambervin inhaled
Drug: Standard of care — The administration of 'StandardTherapy' drugs was done according to the regimen recommended in the 'COVID-19TreatmentGuidelines'(current version)
  Arms: Standard of care

SUMMARY:
This is open-labe randomized multicenter comparative Phase III study conducted in 8 medical facilities. The objective of the study is to assess the efficacy, safety and tolerability of Ambervin for intramuscular and inhaled administration in complex therapy COVID-19 compared with the Standard of care (SOC) in hospitalized patients with moderate COVID-19.

DETAILED DESCRIPTION:
Upon signing the informed consent form and screening, 313 eligible patients hospitalized with COVID-19 were randomized at a 1:1:1 ratio to receive either Ambervin intramuscular 1mg 1 times a day for 10 days or Ambervin inhaled 10mg 1 times a day for 10 days or SOC.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of the Informed Consent Form of thePatient Information Leaflet (PIL) signed and dated bypatient.
2. Men and women aged 18 to 80 years inclusive at thetime of signing the Informed Consent Form in PIL.
3. Confirmed case of COVID-19 at the time ofscreening based on SARS-CoV-2 RNA test usingnucleic acid amplification (NAA) method. It isacceptable to include a patient with a presumptiveCOVID-19 diagnosis prior to receiving the results ofSARS-CoV-2 RNA test made at the screening stage.
4. Hospital admission due to COVID-19.
5. Moderate severity infection with SARS-CoV-2: Clinical signs (the presence of at least 2 of the following criteria):

   * body temperature > 38 °C;
   * RR > 22/min;
   * CT pattern typical of a viral lesion
   * shortness of breath on exertion;
   * SpO2 < 95%;
   * Serum CRP > 10 mg/L.
6. Lesion volume is minimal or moderate; CT 1-2.
7. Patient's consent to use reliable contraceptive methods through out the study and within 1 month for women and 3 months for men after its completion. Reliable means of contraception are: sexualabstinence, use of condom in combination withspermicide.

Women incapable of childbearing may also participate inthe study (with past history of: hysterectomy, tubal ligation,infertility, menopause for more than 2 years), as well asmen with infertility or a history of vasectomy

Exclusion Criteria:

1. Hypersensitivity to components of the study drug.
2. Impossibility of CT procedure (for example, gypsumdressing or metal structures in the field of imaging).
3. Obstacles or inability to perform intramuscular injections and / or inhalations
4. Arterial hypotension (a decrease in blood pressure (BP) below 100/60 mm Hg) at the time of screening and / or a history of hypotensive crises.
5. The need for the use of drugs from the list of prohibited therapies.
6. Availability of criteria for severe and extremely severe disease at the time of screening
7. Presence within 6 months prior to screening of a probable or confirmed case of moderate COVID-19
8. History of presumptive or confirmed COVID-19 caseof moderate, severe and extremely severe course ofthe disease.
9. Vaccination less than 4 weeks prior to screening.
10. The need for treatment in the intensive care unit at the time of screening.
11. Impaired liver function (AST and/or ALT ≥ 2 UNLand/or total bilirubin ≥ 1.5 UNL) at the time ofscreening.
12. Renal impairment (GFR < 60 ml/min) at the time of screening.
13. Positive testing for HIV, syphilis, hepatitis B and/or C.
14. Chronic heart failure FC III-IV according to New York Heart Association (NYHA) functional classification.
15. Malignancies in the past medical history.
16. Alcohol, pharmacological and/or drug addiction in the past medical history and/or at the time of screening.
17. Epilepsy in history.
18. Schizophrenia, schizoaffective disorder, bipolardisorder, or other history of mental pathology orsuspicion of their presence at the time of screening.
19. Severe, decompensated or unstable somatic diseases (any disease or condition that threaten thepatient's life or impair the patient's prognosis, and also make it impossible for him/her to participate in the clinical study).
20. Any history data that the investigating physician believes could lead to complication in the interpretation of the study results or create an additional risk to the patient as a result of his/her participation in the study.
21. Patient's unwillingness or inability to comply with procedures of the Study Protocol (in the opinion of physician investigator).
22. Pregnant or nursing women or women planning pregnancy.
23. Participation in another clinical study for 3 monthsprior to inclusion in the study.
24. Other conditions that, according to the physicianinvestigator, prevent the patient from being includedin the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Prevalence of patients with category 0-1 as per categorical ordinal clinical improvement WHO scale | From baseline to Visit 4 (days 14-15)
  The proportion of patients with category 0-1 as per the categorical ordinal clinical improvement scale

SECONDARY OUTCOMES:
Prevalence of patients with clinical status less than 4 points on the categorical ordinal WHO scale of clinical improvement | From baseline to Visit 3 (days 11-12) and 4 (days 14-15)
  The proportion of patients with clinical status less than 4 points on the categorical ordinal WHO scale of clinical improvement
Frequency of improvement in clinical status on a categorical ordinal WHO scale of clinical improvement of 2 or more categories | From baseline to Visit 3 (days 11-12) and 4 (days 14-15)
  The proportion of patients with clinical status on a categorical ordinal WHO scale of clinical improvement of 2 or more categories
Time to improve clinical status on a categorical ordinal scale of clinical improvement by ≥ 1 point. | From baseline to Visit 6 (study completion, day 28±1)
  Number of days to improve clinical status on a categorical ordinal scale of clinical improvement by ≥ 1 point.
Prevalence of patients eligible for discharge to continue outpatient treatment according to BMR | From baseline to Visit 2 (days 6-7), 3 (days 11-12)
  The proportion of patients eligible for discharge to continue outpatient treatment according to current Cuidelines
Prevalence of patients with RR < 22/min | From baseline to Visit 2 (days 6-7), 3 (days 11-12)
  The proportion of patients with RR < 22/min
Prevalence of patients with CRP level < 10 mg/l | From baseline to Visit 2 (days 6-7), 3 (days 11-12)
  The proportion of patients with CRP level < 10 mg/l
Prevalence of patients with blood lymphocytes > 1.2 x 10(9)/L | From baseline to Visit 2 (days 6-7), 3 (days 11-12)
  The proportion of patients with blood lymphocytes > 1.2 x 10(9)/L
Assessment of the degree of lung damage according to CT | From baseline to Visit 4 (days 14-15)
  The degree of lung damage according to CT
Prevalence of patients with SpO2 ≥ 95% on 2 consecutive days | From baseline to Visit 2 (days 6-7), 3 (days 11-12), 4 (days 14-15)
  The proportion of patients with SpO2 ≥ 95% on 2 consecutive days
The frequency of transfer of patients to the intensive care unit and intensive care | From baseline to Visit 6 (study completion, day 28±1)
  The proportion of patients transferred to the intensive care unit and intensive care
The frequency of cases of the use of high flow oxygen therapy, non-invasive and invasive ventilation of lung, ECMO | From baseline to Visit 6 (study completion, day 28±1)
  The proportion of patients who used high flow oxygen therapy, non-invasive and invasive ventilation of lung, ECMO
The frequency of cases of ARDS | From baseline to Visit 6 (study completion, day 28±1)
  The proportion of patients with ARDS
The frequency of patients with a fatal outcome | From baseline to Visit 6 (study completion, day 28±1)
  The proportion of patients with a fatal outcome

CONTACTS AND LOCATIONS:
Overall Officials: Dmitriy Pushkar, Principal Investigator — Moscow State Clinical Hospital №50
Locations (10):
- Russia (10):
  - Budgetary institution of the Chuvash Republic "Emergency Hospital", Cheboksary
  - City clinical Hospital №24, Moscow
  - Infectious Clinical Hospital No.1, Moscow
  - State Budgetary Healthcare Institution City Clinical Hospital named after S. I. Spasokukotskiy of Moscow Healthcare Department, Moscow
  - Regional Clinical Hospital, Ryazan
  - Ryazan State Medical University named after academician I.P. Pavlov of Ministry of Health of the Russian Federation, Ryazan
  - Ogarev Mordova State University of Ministry of Health of the Russian Federation, Saransk
  - City Hospital No. 40 Kurortny District, Sestroretsk
  - Regional State Budget Healthcare Institution "Clinical hospital No. 1", Smolensk
  - Voronezh Regional Clinical Hospital No.1, Voronezh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] L.A. Balykova, O.A. Radaeva, K.Ya. Zaslavskaya, P.A. Bely, V.F. Pavelkina, N.A. Pyataev, A.Yu. Ivanova, G.V. Rodoman, N.E. Kostina, V.B. Filimonov, E.N. Simakina, D.A. Bystritsky, A.S. Agafina, K.N. Koryanova, D.Yu. Pushkar. Efficacy and safety of original drug based on hexapeptide succinate in complex COVID-19 therapy in adults hospitalized patients. Pharmacy & Pharmacology. 2022;10(6):573-588. DOI: 10.19163/2307-9266-2022-10-6-573-588
- See also: Cyberleninka is an open access scientific electronic library — https://cyberleninka.ru/article/n/effektivnost-i-bezopasnost-originalnogo-preparata-na-osnove-suktsinata-geksapeptida-v-kompleksnoy-terapii-covid-19-u-vzroslyh